CLINICAL TRIAL: NCT01529736
Title: Prospective Randomized-controlled Study of the Integration Success of Osseotite Implants Placed With Different Insertion Procedures
Brief Title: Randomized Study of Integration Success of Osseotite Dental Implants Placed Using Different Insertion Procedures
Acronym: Pegasus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZimVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3004
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Partial Edentulism; Tooth Disease
Keywords: edentulism; dental implants; early loading; crestal bone level; high torque insertion; low torque insertion; randomized; Osseotite; clinical study
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High torque insertion (Experimental): High torque insertion
  Interventions: Procedure: High torque insertion
- Low torque insertion (Active Comparator): Low torque insertion
  Interventions: Procedure: Low torque insertion

INTERVENTIONS:
Procedure: High torque insertion — Osseotite implant placed with high insertion torque forces
  Other Names: Osseotite endosseous dental implant
  Arms: High torque insertion
Procedure: Low torque insertion — Osseotite implant placed with low insertion torque forces
  Other Names: Osseotite endosseous dental implant
  Arms: Low torque insertion

SUMMARY:
Osseotite implants placed with higher insertion torque (TEST procedure) will have higher initial stability and integration success than those placed with lower insertion torque forces.

DETAILED DESCRIPTION:
Osseotite implants will be placed using the standard lower insertion torque forces and compared to implants placed using higher insertion torque forces.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex and older than 18 years of age
* patients needing a minimum of 3 implants to treat partial edentulism
* patients physically able to tolerate surgical and restorative dental procedures
* patients agreeing to all protocol visits

Exclusion Criteria:

* patients with infection or severe inflammation at the intended treatment sites
* patients smoking greater than 10 cigarettes per day
* patients with uncontrolled diabetes mellitus
* patients with uncontrolled metabolic diseases
* patients who received radiation treatment to the head in the past 12 months
* patients needing bone grafting at the intended treatment sites
* patients known to be pregnant at screening visit
* patients with para-functional habits like bruxing and clenching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
primary stability countertorque measures | 4 months
  resistance to countertorque measures showing primary stability success of implants

SECONDARY OUTCOMES:
cumulative success rate | 1 year
  Crestal bone regression (amount of bone loss measured) and equivalence in integration success (implant mobility)

CONTACTS AND LOCATIONS:
Overall Officials: Armando Estefan, DMD, Principal Investigator — Universidad Javeriana
Locations (1):
- Universidad Javeriana, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided